CLINICAL TRIAL: NCT04097145
Title: A Prospective, Multicenter, Randomized, Controlled Pivotal Trial to Evaluate the Safety and Effectiveness of Transcatheter Tricuspid Valve Repair With the Edwards PASCAL Transcatheter Valve Repair System and Optimal Medical Therapy (OMT) Compared to OMT Alone in Patients With Tricuspid Regurgitation
Brief Title: Edwards PASCAL Transcatheter Valve Repair System Pivotal Clinical Trial
Acronym: CLASP II TR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-07
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Tricuspid Regurgitation; Tricuspid Valve Insufficiency; Tricuspid Valve Disease
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Edwards PASCAL System & OMT (Experimental): Transcatheter tricuspid valve repair with the Edwards PASCAL system in patients on optimal medical therapy (OMT) with tricuspid regurgitation
  Interventions: Device: Edwards PASCAL System
- Optimal Medical Therapy (OMT) (Active Comparator): Optimal medical therapy (OMT) alone in patients with tricuspid regurgitation
  Interventions: Drug: Optimal Medical Therapy
- Single-Arm Registry (Experimental): Transcatheter tricuspid valve repair with the Edwards PASCAL System in conjunction with optimal medical therapy (OMT) in patients with tricuspid regurgitation who are not eligible for randomization
  Interventions: Device: Edwards PASCAL System
- Continued Access Study (Experimental): Transcatheter tricuspid valve repair with the Edwards PASCAL system in patients on optimal medical therapy (OMT) with tricuspid regurgitation
  Interventions: Device: Edwards PASCAL System

INTERVENTIONS:
Device: Edwards PASCAL System — Transcatheter tricuspid valve repair with the Edwards PASCAL System in patients on optimal medical therapy
  Other Names: Transcatheter tricuspid valve repair (TTVr)
  Arms: Edwards PASCAL System & OMT
Drug: Optimal Medical Therapy — Optimal Medical Therapy alone in patients with tricuspid regurgitation
  Arms: Optimal Medical Therapy (OMT)
Device: Edwards PASCAL System — Transcatheter tricuspid valve repair with the Edwards PASCAL System in conjunction with OMT
  Arms: Single-Arm Registry
Device: Edwards PASCAL System — Transcatheter tricuspid valve repair with the Edwards PASCAL system in patients on optimal medical therapy (OMT) with tricuspid regurgitation
  Arms: Continued Access Study

SUMMARY:
To establish the safety and effectiveness of the Edwards PASCAL Transcatheter Repair System in patients with symptomatic severe tricuspid regurgitation who have been determined to be at an intermediate or greater estimated risk of mortality with tricuspid valve surgery by the cardiac surgeon with concurrence by the local Heart Team

DETAILED DESCRIPTION:
A Prospective, multicenter, randomized, controlled pivotal trial to evaluate the safety and effectiveness of transcatheter tricuspid valve repair with the Edwards PASCAL Transcatheter Valve Repair System and optimal medical therapy (OMT) compared to OMT alone in patients with tricuspid regurgitation. Patients will be seen for follow-up visits at discharge, 30 days, 3 months, 6 months, and annually through 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen (18) years of age or older
* Despite medical therapy, per the local Heart Team, patient has signs of TR, symptoms from TR, or prior heart failure hospitalization from TR.
* Severe or greater tricuspid regurgitation
* New York Heart Association (NYHA) Class II-IVa or heart failure hospitalization in the prior 12 months
* Patient is at an intermediate or greater estimated risk of mortality with tricuspid valve surgery as determined by the cardiac surgeon with concurrence by the local Heart Team
* Patient is able and willing to give informed consent, follow protocol procedures, and comply with follow-up visit requirements

Exclusion Criteria:

* Tricuspid valve anatomy not evaluable by TTE or TEE
* Tricuspid valve anatomy precludes proper device deployment and function
* Patient with refractory heart failure requiring, advanced intervention (i.e. patient has or will need left ventricular assist device, or transplantation) (ACC/AHA Stage D heart failure)
* Presence of trans-tricuspid pacemaker or defibrillator leads which meet one of the following:

  1. Would prevent proper TR reduction due to interaction of the lead with the leaflets
  2. Were implanted in the RV within the last 90 days prior to the point of enrollment
* Primary non-degenerative tricuspid disease
* Previous tricuspid valve repair or replacement that would interfere with placement of PASCAL
* Clinically significant, untreated coronary artery disease requiring revascularization, unstable angina, evidence of acute coronary syndrome, recent myocardial infarction
* Significant intra-cardiac mass, thrombus, or vegetation per echo core lab assessment
* Deep vein thrombosis (DVT) or pulmonary embolism (PE) in the last 90 days
* Recent Stroke
* Active gastrointestinal (GI) bleeding
* Presence of infiltrative cardiomyopathy or valvulopathy (including carcinoid, amyloidosis, sarcoidosis, hemochromatosis) or significant congenital heart disease, including but not limited to atrial septal defect, RV dysplasia, and arrhythmogenic RV
* Need for emergent or urgent surgery for any reason, any planned cardiac surgery within the next 12 months (365 days), or any planned percutaneous cardiac procedure within the next 90 days
* Any of the following cardiovascular procedures:

  1. Percutaneous coronary, intracardiac, or endovascular intervention within the last 30 days prior to the point of enrollment
  2. Carotid surgery within 30 days prior to the point of enrollment
  3. Direct current cardioversion within the last 30 days prior to the point of enrollment
  4. Leadless RV pacemaker implant within the last 30 days prior to the point of enrollment
  5. Cardiac surgery within 90 days prior to the point of enrollment
* Severe aortic, mitral and/or pulmonic valve stenosis and/or regurgitation
* Known history of untreated severe symptomatic carotid stenosis or asymptomatic carotid stenosis
* Active endocarditis within the last 90 days or infection requiring antibiotic therapy within the last 14 days
* Patient is oxygen-dependent or requires continuous home oxygen
* Pregnant, breastfeeding, or planning pregnancy within the next 12 months (365 days)
* Concurrent medical condition with a life expectancy of less than 12 months in the judgment of the Investigator
* Patient is currently participating in another investigational biologic, drug, or device clinical study
* Patient has other medical, social, or psychological conditions that preclude appropriate consent and follow-up, or the patient is under guardianship
* Any patient considered to be vulnerable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint including all-cause mortality, RVAD implantation or heart transplant, tricuspid valve intervention, heart failure hospitalizations, and Quality of Life improvement (measured by KCCQ score) | 12 months
  Comparison of number of participants with composite endpoint events between experimental and active comparator arms

SECONDARY OUTCOMES:
1 Grade Reduction in TR Severity | 6, 12 months
  Total number of participants with at least 1 grade reduction in TR severity
Quality of Life (QOL) as Measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) | 3, 6, and 12 months
  Change in KCCQ score from baseline
All Cause Mortality | 12 months, 24 months
  Total number of deaths from any cause
Death and Heart Failure Hospitalizations | 12 months
  Total number of deaths and hospital admissions due to heart failure
All-cause Hospitalization | 12 months
  Total number of hospitalizations due to any cause
Right ventricular end-diastolic diameter (RVEDD mid) | 12 months
  Change in right ventricular end-diastolic diameter (RVEDD mid)
Major Adverse Events (MAEs) | 30 days
  Overall rate of Major Adverse Events (MAEs)
Reduction in TR grade | Intraprocedural post-implantation
  Reduction in TR severity as assessed by TEE pre- and post-implantation
All-Cause Mortality | 12 months, annually through 5 years
  Total number of deaths from any cause
Heart failure hospitalizations | 12 months, annually through 5 years
  Total number of hospital admissions due to heart failure
Non-elective tricuspid valve re-intervenitions (percutaneous or surgical) | 12 months, annually through 5 years
  Total number of non-elective tricuspid valve re-interventions
Durable RVAD implantation or heart transplant | 12 months, annually through 5 years
  Total number of patients requiring RVAD impantantion or heart transplant
Need for paracentesis | 12 months, annually through 5 years
  Total nunber of patients who required paracentesis
All cause mortality or the first heart failure hospitalization for patients with massive or torrential TR at baseline | 12, 24 months
  Time to death or first heart failure hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Martin B. Leon, MD, Principal Investigator — Columbia University; Michael J. Mack, MD, Principal Investigator — Baylor Scott and White Health; Charles Davidson, MD, Principal Investigator — Northwestern University; Allen Anderson, MD, Study Chair — UT Health San Antonio; Gorav Ailawadi, MD, Study Chair — University of Michigan
Locations (79):
- United States (73):
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Tucson Medical Center Healthcare, Tucson, Arizona
  - University of California, Irvine, Irvine, California
  - SCPMG - Kaiser San Diego, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - St. Joseph Hospital, Denver, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - The Cardiac and Vascular Institute Research Foundation, Gainesville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - NCH Healthcare System, Naples, Florida
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Emory University Hospital Midtown / Emory University - St. Joseph's Hospital, Atlanta, Georgia
  - Piedmont Healthcare, Inc., Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Ascension St. Vincent Heart Center Cardiovascular Research Institute, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Ochsner Medical Center, New Orleans, Louisiana
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - St. Mary's of Ascension Research, Saginaw, Michigan
  - Fairview Health Services, Maplewood, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Providence St. Patrick Hospital, Missoula, Montana
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Health Systems, Camden, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - State University of New York at Buffalo, Buffalo, New York
  - Columbia University Irving Medical Center/NYPH, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Lenox Hill Hospital, Northwell Health /Northshore University Hospital Manhasset, New York, New York
  - Rochester General Hospital, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - Montefiore Medical Center / Arts Pavilion / Hutchinson Metro Center Clinic / Weiler Hospital / Moses Hospital, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - The Christ Hospital, Cincinnati, Ohio
  - TriHealth-Bethesda North Hospital, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Oklahoma Heart Institute at Hillcrest Medical Center, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Hershey, Hershey, Pennsylvania
  - Pennsylvania Presbyterian Medical Center / Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pinnacle Health Cardiovascular Institute/UPMC Pinnacle, Wormleysburg, Pennsylvania
  - Lankenau Heart Institute, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Erlanger Health System, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - HCA Houston Healthcare Medical Center, Houston, Texas
  - Baylor College of Medicine St. Luke's Medical Center, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - UTHealth/Memorial Hermann Hospital, Houston, Texas
  - Baylor Scott & White - The Heart Hospital - Plano, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
  - St. George Regional Hospital, St. George, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Carilion Medical Center, Roanoke, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (6):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Hamilton Health Services, Hamilton, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No